CLINICAL TRIAL: NCT02888184
Title: Neuron Specific Enolase and Glasgow Motor Score Remain Useful Tools for Assessing Neurological Prognosis After Out-of-hospital Cardiac Arrest Treated With Therapeutic Hypothermia
Brief Title: Identification of Neurological Prognostic Markers of Cardiac Arrest Patients Alive on 3rd Day
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: IRB 14 01 01
Record Dates: First submitted 2016-08-30; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
The aim of the study is to identify prognostication predictors of 6-months neurological outcome in survivors at day 3 after cardiac arrest (CA) treated with therapeutic hypothermia (TH).

DETAILED DESCRIPTION:
Cardiac arrest (CA) management remains challenging. As fewer than 20% of patients survive to discharge, early prognostication of functional outcome needs accurate prediction.Survivors outcome depends on initial CA conditions (cause, duration and severity of ischemic injury) that may lead to the post-cardiac arrest syndrome, associated with high mortality. Hypoxic-ischemic encephalopathy is the second cause of poor outcome after CA. Indeed, most survivors remain comatose or in a vegetative state leading to decisions to withdraw life support. Thus, the American Academy of Neurology had proposed a decision algorithm for use in prognostication of comatose survivors published in 2006.Before the widespread use of therapeutic hypothermia (TH), predictor factors of neurological outcome were: serum neuron-specific enolase (NSE), N20 somatosensory-evoked potentials (SSEP), status epilepticus, pupil and corneal reflexes and Glasgow coma score motor response (GCS-M). Therapeutic hypothermia is recommended in the management of CA.It has been associated with improved outcome after ventricular fibrillation out-of-hospital cardiac arrest (OHCA). However, TH may interfere with clinical examination and electrophysiological predictors (EEG, SSEP) making prognostication of functional outcome hardiest.The use of sedative drugs and muscle paralysis during TH is another cause of delayed neurological assessment and prognostication.The NSE cutoff values to predict poor neurological outcome are not well defined and can be influenced by TH either.The present study aims at identifying clinical, electrophysiological and biological prognostication predictors of 6-month neurological outcome in survivors at day 3 after CA treated by TH. Neurological functional status was assessed using the 5-item scale Cerebral Performance Category (CPC). Neurological status was retrospectively assessed at 6 months: CPC of 1 or 2 was defined as good neurological outcome and CPC of 3 to 5 were defined as poor neurological outcome. Deaths in the first 3 days and decisions to withdraw or to withhold life support were also collected. The following prognostication factors were tested: neurological examination at day 3 and 7 including corneal and pupillary reflexes, GCS-M, status epilepticus, electro-encephalogram (EEG), SSEPs and NSE levels between day 2 and day 3.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* successfully resuscitated of out-of-hospital cardiac arrest (OHCA)
* patients admitted to ICU

Exclusion Criteria:

* in-hospital cardiac arrest patients
* death before ICU admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients (≥ 18 years) successfully resuscitated of out-of-hospital cardiac arrest (OHCA) and admitted to ICU.
Sampling Method: Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2010-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Neurological functional status assessed by the 5-item scale Cerebral Performance Category (CPC) at 6 months. | 6 month